CLINICAL TRIAL: NCT07044167
Title: Development of a Novel Polyphenol-Enriched Functional Product for the Treatment of Overweight and Obesity
Brief Title: Innovative Functional Product for Overweight and Obesity
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Carmen Lucas Abellán (Other)
Collaborators: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Sponsor-Investigator, Carmen Lucas Abellán, Principal Investigator, Universidad Católica San Antonio de Murcia
Organization: Universidad Católica San Antonio de Murcia (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CE112402
Record Dates: First submitted 2025-05-20; First posted 2025-06-29 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Obesity and Overweight; Overweight or Obese; Overweight or Obese Adults; Obese Subjects; Overweight/Obesity
Keywords: Obesity; Overweight; Polyphenols; Functional food; Randomized controlled trial; Metabolic health
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Daily consumption of the polyphenol-enriched functional product for 60 days.
  Interventions: Dietary Supplement: Polyphenol-enriched functional product
- Control (Placebo Comparator): Identically appearing placebo capsules consumed for 60 days.
  Interventions: Dietary Supplement: Control without active polyphenols

INTERVENTIONS:
Dietary Supplement: Polyphenol-enriched functional product — Polyphenol-enriched functional product
  Arms: Experimental
Dietary Supplement: Control without active polyphenols — Product with identical characteristics to the experimental product, but without active polyphenols.
  Arms: Control

SUMMARY:
The aim of this randomized, parallel, two-arm, placebo-controlled, quadruple-blind clinical trial is to evaluate the efficacy of a polyphenol-enriched functional product in individuals with overweight or obesity, focusing primarily on body composition, insulin sensitivity, inflammatory markers, and other metabolic health parameters.

DETAILED DESCRIPTION:
The duration of the study will be 60 days during which the investigational product or placebo will be consumed daily according to the assignment.

Subjects will be randomized to each of the study arms (consumption of the polyphenol-enriched product or control product).

ELIGIBILITY:
Inclusion Criteria:

* Individuals of both sexes, aged 18 years or older.
* Body Mass Index (BMI) between 25 and 35.
* Clinical diagnosis of overweight or obesity according to established criteria.
* Ability to understand and sign the informed consent form.

Exclusion Criteria:

* Presence of severe or terminal chronic diseases.
* Current treatment with antioxidants or similar dietary supplements.
* Known allergies to any of the product components.
* Pregnancy or breastfeeding.
* Participation in another clinical trial within the past 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in Body Weight | Day 1 and Day 60
  Evaluation of differences in body weight (kg)
Change in fat mass | Day 1 and Day 60
  Evaluation of differences in fat mass (kg)
Change in fat mass (%) | Day 1 and Day 60
  Evaluation of differences in fat mass percentage (%)
Change in Body Mass Index (BMI) | Day 1 and Day 60
  BMI will be calculated from measured weight and height using the formula weight (kg) / height² (m²).

SECONDARY OUTCOMES:
Change in fasting glucose | Day 1 and Day 60.
  Assessment of changes in fasting glucose levels (mg/dL)
Change in fasting insulin | Day 1 and Day 60.
  Assessment of changes in insulin levels.
Change in plasma leptin levels | Day 1 and Day 60
  Leptin levels will be measured in fasting plasma samples using ELISA at baseline and after the intervention (pg/mL).
Change in plasma ghrelin levels | Day 1 and Day 60
  Ghrelin levels will be measured in fasting plasma samples using ELISA at baseline and after the intervention (ng/mL).
Change in plasma adiponectin levels | Day 1 and Day 60
  Adiponectin levels will be measured in fasting plasma samples using ELISA at baseline and after the intervention (ng/mL).
Change in plasma SOCS3 levels | Day 1 and Day 60
  SOCS3 levels will be measured in fasting plasma samples using ELISA at baseline and after the intervention (pg/mL).
Change in plasma interleukin-1 (IL-1β) levels | Day 1 and Day 60
  Interleukin-1 (IL-1β) levels will be measured in fasting plasma samples using ELISA at baseline and after the intervention (pg/mL).
Change in plasma interleukin-6 (IL-6) levels | Day 1 and Day 60
  Interleukin-6 (IL-6) levels will be measured in fasting plasma samples using ELISA at baseline and after the intervention (pg/mL).
Change in plasma interleukin-10 (IL-10) levels | Day 1 and Day 60
  Interleukin-10 (IL-10) levels will be measured in fasting plasma samples using ELISA at baseline and after the intervention (pg/mL).
Change in plasma oxidized LDL (oxLDL) levels | Day 1 and Day 60
  Oxidized LDL (oxLDL) levels will be measured in fasting plasma samples using ELISA at baseline and after the intervention (pg/mL).
Change in plasma malondialdehyde (MDA) levels | Day 1 and Day 60
  Malondialdehyde (MDA) levels will be measured in fasting plasma samples using ELISA at baseline and after the intervention (ng/mL).
Change in plasma superoxide dismutase (SOD) levels | Day 1 and Day 60
  superoxide dismutase (SOD) levels will be measured in fasting plasma samples using ELISA at baseline and after the intervention (pg/mL).
Changes in C-reactive protein (CRP) | Day 1 and Day 60
  Measurement of changes in C-reactive protein (mg/L)

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Lucas Abellán, Principal Investigator — Universidad Católica San Antonio de Murcia
Locations (1):
- UCAM San Antonio Catholic University of Murcia, Murcia, Murcia 30107, Murcia, Spain